CLINICAL TRIAL: NCT01634061
Title: Phase Ib Dose Finding Study of Abiraterone Acetate Plus BEZ235 or BKM120 in Patients With Castration-resistant Prostate Cancer.
Brief Title: Phase Ib of Abiraterone Acetate Plus BEZ235 or BKM120 in Castration-resistant Prostate Cancer (CRPC) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235D2101; 2012-002250-23 (EudraCT Number)
Record Dates: First submitted 2012-06-26; First posted 2012-07-06 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2015-09

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Castration-resistant prostate cancer, abiraterone acetate, BEZ235, BKM120, dose escalation, abiraterone acetate failure
MeSH Terms: interventions — dactolisib; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose escalation: BEZ235 + Zytiga® (Experimental): BEZ235 oral twice daily: 200 mg, 300 mg, and 400 mg dose levels to be tested in the dose escalation part in combination with abiraterone acetate Zytiga® abiraterone acetate oral once daily: 1000 mg taken with low dose prednisone as per the label
  Interventions: Drug: BEZ235
- Dose escalation: BKM120 + Zytiga® (Experimental): BKM120 oral once daily: 60 mg, 80 mg and 100 mg dose levels to be tested in the dose escalation part in combination with abiraterone acetate Zytiga® abiraterone acetate oral once daily: 1000 mg taken with low dose prednisone as per the label
  Interventions: Drug: BKM120
- Dose expansion: BEZ235 + Zytiga® (Experimental): BEZ235 oral twice daily: 200 mg, 300 mg, and 400 mg dose levels to be tested in the dose escalation part in combination with abiraterone acetate
  Zytiga® abiraterone acetate oral once daily: 1000 mg taken with low dose prednisone as per the label
  Interventions: Drug: BEZ235
- Dose Expansion: BKM120 + Zytiga® (Experimental): BKM120 oral once daily: 60 mg, 80 mg and 100 mg dose levels to be tested in the dose escalation part in combination with abiraterone acetate Zytiga® abiraterone acetate oral once daily: 1000 mg taken with low dose prednisone as per the label
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BEZ235 — BEZ235 will be supplied as 50mg, 100mg, 200mg, 300mg and 400mg SDS sachets. At each patient's visit, patient will reecive a prescription of an adequate drug supply for self administration at home.
  Arms: Dose escalation: BEZ235 + Zytiga®
Drug: BKM120 — BKM120 will be supplied as 10mg and 50mg hard gelatin capsules. At each patient's visit, patient will reecive a prescription of an adequate drug supply for self administration at home.
  Arms: Dose escalation: BKM120 + Zytiga®
Drug: BEZ235 — BEZ235 will be supplied as 50mg, 100mg, 200mg, 300mg and 400mg SDS sachets. At each patient's visit, patient will reecive a prescription of an adequate drug supply for self administration at home.
  Arms: Dose expansion: BEZ235 + Zytiga®
Drug: BKM120 — BKM120 will be supplied as 10mg and 50mg hard gelatin capsules. At each patient's visit, patient will reecive a prescription of an adequate drug supply for self administration at home.
  Arms: Dose Expansion: BKM120 + Zytiga®

SUMMARY:
This is an open label study of abiraterone acetate in combination with BEZ235 and abiraterone acetate in combination with BKM120 in CRPC patients with abiraterone acetate failure.

DETAILED DESCRIPTION:
A dose-escalation part will first determine the maximum tolerated dose (MTD) and/or recomended dose for expansion (RDE) of abiraterone acetate in combination with BEZ235 and abiraterone acetate in combination with BKM120 in CRPC patients with abiraterone acetate failure.

Subsequently, the MTD and/or RDE of each combination will be investigated in two expansion treatment groups of CRPC patients who have failed abiraterone acetate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult males ≥ 18 years old
* Eastern Cooperative Oncology Group Performance Status ≤ 2
* Patient must have a castrate level of testosterone (<= 50 ng/dL or 1.7 nmol/L). ( Castrate status must be maintained by continued GnRH analogues unless patient has undergone surgical orchiectomy).
* Histologically or cytologically confirmed diagnosis of advanced or metastatic prostate cancer.
* Advanced or metastatic castration-resistant prostate cancer progression after abiraterone acetate failure
* Patients should have no more than 2 lines of prior chemotherapies including cytotoxic agents
* Discontinuation of all anti-androgen, anti-neoplastic or investigational treatment >= 4 weeks (6 weeks for bicalutamide).

Exclusion Criteria:

* Previous treatment with PI3K pathway inhibitors (e.g. PI3K, AKT, mTOR inhibitor), ketoconazole, CYP17 inhibitors (exception of AA), or enzalutamide.
* Patient has active uncontrolled or symptomatic CNS metastases
* Inadequately controlled hypertension (e.g. systolic blood pressure >=160 mmHg or diastolic blood pressure >=95 mmHg)
* Patient has a QTcF > 480 msec on the screening ECG (using the QTcF formula), has a short/long QT syndrome, or history of QT prolongation/Torsades de Pointes
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others)
* Patients who experienced dose reductions and/or treatment interruptions due to abiraterone acetate related toxicities (i.e. serious AEs, AEs, liver toxicities during abiraterone acetate treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | from days 1-35 in BEZ235/abiraterone acetate arm and from days 1-28 in BKM120/abiraterone acetate arm
  Dose escalation part: Determine MTD and /or RDE of the combinations abiraterone acetate + BEZ235 and abiraterone acetate + BKM120 by assessing the incidence of DLTs in cycle 1
Prostate specific antigen (PSA) decline ≥ 30% | At week 12 or later after treatment discontinuation
  Dose expansion part: Assess anti-tumor activity of the combinations (abiraterone acetate + BEZ235 and abiraterone acetate + BKM120) in castration-resistant prostate cancer patients with abiraterone acetate failure as on treatment PSA progression according to prostate cancer working group criteria 2 (PCWG2) by assessing PSA decline ≥ 30% at Week 12 or later.

SECONDARY OUTCOMES:
Number of patients with at least one adverse event | Treatment start until 30 days after the last dose
radiological Progression Free Survival as per RECIST 1.1 and PCWG2 | Every 12 weeks until disease progression
radiological Response Rate according to RECIST 1.1 | Every 12 weeks until disease progression
Overall Survival | From treatment start until 75% of deaths from any cause have occurred
Number and percentage of patients with laboratory abnormalities | Treatment start until 30 days after the last dose
Changes in ECG (electrocardiogram) | Treatment start until 30 days after the last dose
Changes in vital signs | Treatment start until 30 days after the last dose
Changes in mood scales | Treatment start until 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (2):
  - Cedars Sinai Medical Center SC, Los Angeles, California
  - Hackensack University Medical Center Hackensack Univ, Hackensack, New Jersey
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Wilrijk
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- France (2):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Villejuif
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Sutton, United Kingdom

REFERENCES:
- See also: Results for CBEZ235D2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15047